CLINICAL TRIAL: NCT01903746
Title: Epidemiology of Septic Shock in Medical or Polyvalent ICU in the North-East Region of France
Status: Terminated | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Quenot PHRC IR 2008
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Severe Sepsis; Persistent Hypotension
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients in septic shock

SUMMARY:
The epidemiology of this study aims and outcome of patients with septic shock in the intensive care unit (or versatile) of the North-East region in france as well as the modalities of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients in septic shock defined by hypotension that is not reversed by volume resuscitation and requires the use of vasopressors.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in septic shock
Sampling Method: Non-Probability Sample
Enrollment: 1495 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Sequential Organ Failure Assessment | baseline

CONTACTS AND LOCATIONS:
Overall Officials: jean pierre Quenot, Principal Investigator — department Medical Intensive Care